CLINICAL TRIAL: NCT01832116
Title: 89Zr-MMOT0530A PET Imaging in Patients With Unresectable Pancreatic or Platinum-resistant Ovarian Cancer Before Treatment With DMOT4039A. A Separate Study to the Phase I Study Protocol DMO4993g
Brief Title: 89Zr-MMOT PET Imaging in Pancreatic and Ovarian Cancer Patients
Acronym: MMOT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMOT imaging
Record Dates: First submitted 2013-04-02; First posted 2013-04-15 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Neoplasms; Ovarian Diseases; Adnexal Diseases; Pancreatic Neoplasms; Digestive System Neoplasms; Digestive System Diseases; Pancreatic Diseases
Keywords: Pancreatic cancer; Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Diseases; Adnexal Diseases; Pancreatic Neoplasms; Digestive System Neoplasms; Digestive System Diseases; Pancreatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tracerinjection (Experimental): Injection of 89Zr-MMOT0530A followed by 2 or 3 PET scans at different time points
  Interventions: Drug: 89Zr-MMOT0530A

INTERVENTIONS:
Drug: 89Zr-MMOT0530A — Injection of 89Zr-MMOT0530A followed by 2 or 3 PET scans at different time points
  Other Names: MMOT

SUMMARY:
The purpose of this multicenter imaging sub study is to evaluate the biodistribution and organ pharmacokinetics of 89Zr-MMOT0530A in patients with unresectable pancreatic or platinum-resistant ovarian cancer. MMOT0530A is a monoclonal antibody that targets an antigen overexpressed in pancreatic and ovarian cancer. Subsequent to imaging with 89Zr-MMOT0530A, patients will be treated with DMOT4039A in the DMO4993g protocol (clinicaltrials.gov identifier NCT01469793) after this study. DMOT4039A is an antibody-drug conjugate composed of the monoclonal antibody MMOT0530A and the mitotic agent monomethyl auristatin (MMAE). By imaging patients with the monoclonal antibody MMOT0530A before treatment, the correlation between tumor uptake of 89Zr-MMOT0530A and response to DMOT4039A therapy will be assessed.

DETAILED DESCRIPTION:
A challenge in current drug development using molecular targeted therapies is the high level of heterogeneity that is present in specific tumor types. The ability to safely and accurately predict the presence or absence of the target is essential for the therapeutic effect of the newly developed drugs. DMOT0439A is one of those novel designed molecular targeted drugs; an antibody-drug conjugate composed of the monoclonal antibody MMOT0530A and the mitotic agent monomethyl auristatin (MMAE). In the DMO4993g protocol (clinicaltrials.gov identifier NCT01469793), the safety and efficacy of DMOT4039A is assessed in patients with unresectable pancreatic or platinum-resistant ovarian cancer. By performing a 89Zr-MMOT0530A PET scan prior to treatment with DMOT4039A, the uptake of the tracer in the primary and metastatic tumor lesions can be evaluated. This is likely to provide important information about target expression, whole body drug distribution and the correlation between tumor uptake and response to therapy. Ultimately the use of a 89Zr- MMOT0530A PET as a complimentary tool for patient selection and risk stratification can be evaluated. In part A of this study, the optimal tracer dose of 89Zr- MMOT0530A and schedule for PET imaging will be determined. In part B patients will have PET imaging before treatment in the DMO4993g study on the dose and time points as assessed in part A.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Histologically documented, incurable, locally advanced or metastatic disease for which no standard therapy exists, consisting of one of the following: Unresectable pancreatic ductal adenocarcinoma or platinum-resistant ovarian cancer
* Measureable disease, defined as at least one bi-dimensionally measurable non-lymph node lesion >/= 1 cm in long-axis diameter on spiral CT scan or at least one bi-dimensionally measurable lymph node measuring >/= 1.5 cm in short-axis diameter on spiral CT scan
* Adequate hematological, renal and liver function

Exclusion criteria:

* Treatment with anti-tumor therapy, including chemotherapy, biologic, experimental or hormonal therapy, within 4 weeks prior to Day 1
* Known active infection
* Current Grade >/= 2 toxicity (except for alopecia, anorexia and fatigue) from prior therapy or Grade >/= 2 neuropathy
* Untreated or active cerebral nervous system (CNS) metastases
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The in vivo biodistribution measured in SUV values and organ pharmacokinetics (PK) of 89Zr-MMOT0530A | Approximately 1 year
  * The accumulation, distribution and localization of 89Zr-MMOT0530A in tumor tissue, organs and blood circulation, as assessed by PET.
  * The quantitative uptake of 89Zr-MMOT0530A expressed in SUV (Standardized Uptake value).

SECONDARY OUTCOMES:
The 89Zr-MMOT0530A tumor uptake measured in SUV related to the response to DMOT4039A therapy according to RECISt 1.1 criteria | Approximately 1 year
  The correlation between the 89Zr-MMOT0530A tumor uptake and response to therapy by performing an 89Zr-MMOT0530A PET scan before DMOT4039A therapy, related to CT/MRI response according to RECIST 1.1 criteria.
Number of patients with adverse events after 89Zr-MMOT0530A injection as a measure of safety and tolerability | Approximately 1 year
  Safety will be assessed by evaluation of incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth G. de Vries, MD PhD, Principal Investigator — University Medical Center Groningen; Henk M Verheul, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - VU Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen